CLINICAL TRIAL: NCT00246168
Title: ULTRACET (Tramadol Hydrochloride and Acetaminophen) add-on Therapy for the Treatment of the Pain of Rheumatoid Arthritis: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: ULTRACET (Tramadol Hydrochloride and Acetaminophen) for the Treatment of Rheumatoid Arthritis Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005929
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; NSAID add-on therapy; tramadol; acetaminophen
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultracet

INTERVENTIONS:
Drug: tramadol hydrochloride + acetaminophen

SUMMARY:
The purpose of this study is to assess the effectiveness of ULTRACETÂ® (a combination analgesic) as add-on therapy in rheumatoid arthritis patients taking an NSAID (e.g. AdvilÂ®, MotrinÂ® or other nonsteroidal anti-inflammatory drug) or a COX-2 inhibitor (e.g. CelebrexÂ®).

DETAILED DESCRIPTION:
This is a randomized, multicenter, placebo-controlled, double-blind study to evaluate the efficacy and safety of ULTRACET® (tramadol 37.5 mg and acetaminophen 325 mg) as add-on therapy in rheumatoid arthritis patients taking an NSAID or a COX-2 inhibitor. The patients will be randomized into 2 treatment groups: The first group will receive one ULTRACET® tablet 3 times per day for 7 days. The second group will receive one placebo tablet 3 times per day for 7 days. The primary efficacy measurement will be the patients' average daily pain score. Safety will be monitored throughout the study. The study hypothesis is that ULTRACET® will be well tolerated and the average daily pain relief score for the ULTRACET® treatment group will be better than that of placebo group. Patients will take one ULTRACET® tablet or placebo by mouth 3 times per day, for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis at least 6 months before the participation in the clinical trial, (defined by having more than 4 of the diagnosis criteria suggested by American College of Rheumatology (ACR
* 1987))
* have been on a stable daily dose of an NSAID or a COX-2 inhibitor for at least 30 days prior to the start of the study
* have arthralgia (arthritis pain in the joints) for at least 2 days before the entering clinical trial, with a pain score on the Visual Analogue Scale (VAS) of 40 mm or greater.

Exclusion Criteria:

* Have had an inadequate response to Tramadol HCl therapy, or have discontinued Tramadol HCl therapy due to adverse events
* have taken Tramadol HCl within 30 days prior to study entry
* have recently taken other medications for pain relief, (other than their daily NSAID or COX-2 inhibitor
* daily use of aspirin at a dose greater than 100 mg per day.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Average daily pain relief score

SECONDARY OUTCOMES:
Average daily pain intensity score; average pain relief and intensity score for the final visit; patient's assessment of physical function; overall assessment by the patient; overall assessment by the investigator; and an evaluation of safety

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.